CLINICAL TRIAL: NCT02847871
Title: Prevention of Loss of Mobility From a Care Pathway Focused on Exercise and Nutrition in Elderly Patients Over 70 Years, in Primary Care. Cluster Randomized Controlled Trial
Brief Title: Elderly Patient at Risk of Loss of Mobility, Exercise - Primary Care, Prevention, Care Pathways
Acronym: PRISME-3P
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 69HCL16_0132
Record Dates: First submitted 2016-07-21; First posted 2016-07-28 (Estimated); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Elderly Patient (>70 Years); Loss of Mobility
Keywords: mobility; exercise; nutrition; primary care; prevention; care pathway; elderly patient
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Multimodal Intervention (Other): The multimodal intervention on mobility will consist of the implementation of a care pathway dedicated in primary care. It will include awareness and training of general practitioners for easy identification, a care associating a dedicated geriatric consultation to rule out underlying pathology, teaching exercises by MAPA (+/- taken care in the presence of MAPA) and nutritional counseling by a dietician. Close collaboration between general practitioners, geriatrician, MAPA and dietician will be established.
  Interventions: Behavioral: PRISME-3P program
- Non interventional (No Intervention): Patients received treatment as part of their standard care: at the discretion of the general practitioner patients

INTERVENTIONS:
Behavioral: PRISME-3P program — PRISM-3P program will consist on a visit in the geriatric centre:
  * Consultation with the geriatrician to rule a condition associated with loss of mobility and not known until now.
  * Perform a nutritional assessment by a dietician followed by appropriate care management.
  * Educational activity based on exercises and physical activity and balance: MAPA teaches exercises to develop strength and balance; gives tips to increase time spent on non-sedentary activities and enhance endurance followed by a monthly phone coaching.
  * At 3 months, in case of no improvement of the SPPB score of 1 point, a training of 10 weeks with two sessions per week will be perform by the MAPA individually or in small patients groups;
  * Implementation of a information exchange processing (mail, phone and book binding) between the various stakeholders.
  Arms: Multimodal Intervention

SUMMARY:
Loss of mobility is predictive of a loss of autonomy and is often the first sign of functional decline. Loss of mobility is also associated with poor perceived quality of life, depressive symptoms, high risk of adverse events such as falls and fractures, to an increased risk to input in institution and mortality's increase.

Consequences and frequency of loss of mobility make essential its identification, evaluation and the practice of preventive measures in primary care.

The implementation of effective interventions in primary care to prevent or delay the loss of mobility is a public health priority.

PRISME-3P program aims to develop and evaluate a dedicated care pathway, in primary care, based on a personalized multimodal intervention: screening, support combining physician, teaching exercises by a specialized Monitor in Adapted Physical Activities (MAPA) and nutritional counseling.

ELIGIBILITY:
Inclusion Criteria:

* Aged > 70 years
* With at least 2 of the following signs:

  1. Difficulty in carrying a shopping bag (load about 4.5 Kg)
  2. Difficulty in getting up from a chair without using arms
  3. Difficulty in climbing 10 stairs
  4. Difficulty in moving, walking slow
  5. Difficulty in walking more than 400 meters without stop
  6. Running time <1 hour / week
  7. Fatigue at modest physical effort: shopping, housework ...
  8. At least two falls in the last year
  9. Weight loss ≥5% in 1 month or weight loss ≥10% in 6 months
* Short Physical Performance Battery score < 10

Exclusion Criteria:

* Locomotor disability not allowing implementation of the protocol according to the investigator
* Life expectancy less than 6 months
* Severe chronic progressive pathologies incompatible with the completion of the physical activity program
* Patient institutionalized in nursing homes
* Advanced Cognitive impairment (MMSE <20)

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 39 (Actual)
Dates: Start 2018-05-16 (Actual); Primary Completion 2021-03-01 (Actual); Study Completion 2021-03-01 (Actual)

PRIMARY OUTCOMES:
Change in Short Physical Performance Battery (SPPB) score | from baseline at 6 months
  Consists in estimating three components: 1. walking, 2. muscular strength and endurance, and 3. balance through short physical exercises (walk on a defined distance, get up from a chair, keep a position up). A score from 1 to 3 for each of the components marks a very low feature of lower limbs. This feature is considered low of 4 in 6, moderated by 7 in 9 and high of 10 in 12.

SECONDARY OUTCOMES:
Evolution of the Short Physical Performance Battery (SPPB) score | Baseline, 3 months (for interventional arm), 6 months and 12 months
  Consists in estimating three components: 1.walking, 2.muscular strength and endurance, and 3. balance through short physical exercises (walk on a defined distance, get up from a chair, keep a position up). A score from 1 to 3 for each of the components marks a very low feature of lower limbs. This feature is considered low of 4 in 6, moderated by 7 in 9 and high of 10 in 12.
Assessment of functional disability by questionnaires | Baseline, 6 months and 12 months
  Functional disability refers to limitations in performing in dependent living tasks, which are often further divided into activities of daily living (ADLs), which include basic activities of hygiene and personal care, and instrumental activities of daily living (IADLs), which include basic activities necessary to reside in the community, such as shopping, managing finances, housekeeping, and meal preparation
Assessment of Quality of Life by questionnaire | baseline, 6 months and 12 months
  The Quality of Life is assessed with the 12-Item Short Form Health Survey (SF-12). The SF-12 is a multipurpose short form survey with 12 questions which were combined, scored, and weighted to create two scales that provide glimpses into mental and physical functioning and overall health-related-quality of life
Number of falls | Baseline, 6 months and 12 months
  Data will be collected by the geriatrician from the patient's medical records
Number of hospitalization | Baseline, 6 months and 12 months
  Data will be collected by the geriatrician from the patient's medical records
Assessment of the Physical Activity by questionnaire | baseline, 6 months and 12 months
  Using the Physical Activity Scale for the Elderly (PASE) auto-questionnaire which is designed to assess the duration, frequency, exertion level, and amount of physical activity undertaken over a seven day period.
Assessment of sedentary time by questionnaire | baseline, 6 months and 12 months
  Using self-report sedentary behavior questionnaire based on the Gardiner questionnaire to assess time spent in behaviors common among older adults: watching television, computer use, reading, socializing, transport and hobbies, and a summary measure (total sedentary time)
Assessment of weight loss | baseline, 6 months and 12 months
  weight in kilograms
Body Mass Index (BMI) | baseline, 6 months and 12 months
  calculating the BMI in kg/m^2
Assessment of nutritional status using MNA scale | baseline, 3 months (for interventional arm depending on the SPPB score), 6 months and 12 months
  Using the Mini Nutritional Assessment (MNA) scale which consists of 18 point-weighted questions in four categories, i.e., anthropometry, global and dietary issues, and self-assessment.
Rate of study participation | Baseline
Monitoring of detailed physical activity performed by patients with diaries outlining the exercise sessions . | at the end of the multimodal intervention (3 months)
  Patient adherence to the multimodal intervention. Monitoring of detailed physical activity performed by patients. Patients were also asked to complete diaries outlining the exercise sessions.
Monitoring of detailed physical activity performed by patients with MAPA assessment. | at the end of the multimodal intervention (3 months)
  Patient adherence to the multimodal intervention. Monitoring of detailed physical activity performed by patients. Patients MAPA assessment.
Rate of compliant General practitioners (GP) associated to the study | at 12 months
Assessment of psychological factors using GDS-4 scale associated with a loss of mobility | baseline, 6 and 12 months
  Using a short Geriatric Depression Scale (GDS-4). The GDS may be used with healthy, medically ill and mild to moderately cognitively impaired older adults.
Assessment of social factors associated with a loss of mobility | baseline
  Using the Evaluation of Precarity and Inequalities in Health Examination Centers (EPICES) score which is related to several socioeconomic indicators (occupation, education, and employment status), to health-related behaviors (smoking and health care use), and morbidity (self-perceived health, dental health, obesity, and diabetes).
Assessment of comorbidities using the index of Charlson | baseline
  Using the index of Charlson which included a closed list of 19 diseases, grouped into 4 subgroups different weighting.
Description of concomitant medications | baseline
  List of active drugs and psychotropic
Type of diagnoses for unknown diseases following the dedicated geriatric consultation. | baseline
  Description of pathologies possibly associated with a symptomatic loss of mobility.
Percentage of diagnoses for unknown diseases following the dedicated geriatric consultation. | baseline
  Description of pathologies possibly associated with a symptomatic loss of mobility.

CONTACTS AND LOCATIONS:
Overall Officials: Marc BONNEFOY, Pr, Principal Investigator — Hospices Civils de Lyon
Locations (1):
- Service de Médecine Gériatrique. Groupement Hospitalier Sud. Hospices Civils de Lyon., Pierre-Bénite, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Perrotin S, Gilbert T, Dupuis M, Villeneuve L, Bin-Dorel S, Klich A, Letrilliart L, Bonnefoy M. A multimodal and multidisciplinary program to prevent loss of mobility in patients aged over 70 years: study protocol of a multicenter cluster randomized study in primary care (the PRISME-3P study). BMC Geriatr. 2019 Feb 19;19(1):48. doi: 10.1186/s12877-019-1059-5. PMID 30782118